CLINICAL TRIAL: NCT07060274
Title: Halo Sign Vanishing Time After Steroids Outbreak in GCA Patients
Acronym: Halo-A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHM-2025/S06/02
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Giant Cell Arteritis (GCA); Doppler Ultrasound
Keywords: Giant cell arteritis; echo-Doppler; Doppler ultrasonography; Halo sign; steroids
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Intervention Model Description: A single group is followed during 15 days with steroids treatment and the time until the halo disappears is monitored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Timeframe for Halo sign resolution on Doppler ultrasound (Experimental): Doppler ultrasound of temporal arteries at D0, D3 and D7 (+/- D15) after initiation of corticosteroid therapy.
  Interventions: Procedure: Doppler Ultrasound

INTERVENTIONS:
Procedure: Doppler Ultrasound — Doppler ultrasound of temporal arteries at D0, D3 and D7 (+ D15 if halo detected at D7) after initiation of corticosteroid therapy.

SUMMARY:
Giant cell arteritis (GCA) is a rare disease characterized by vasculitis of the large arterial trunks targeting the thoracic aorta and its dividing branches, affecting adults over the age of 50. Vasculitis lesions cause thickening of the arterial wall, visible on temporal artery biopsy (TAB) or vascular imaging (echo-Doppler, angio-CT, angio-MRI, 18FDG PET-CT). This is a severe disease that can lead to blindness. Early diagnosis is essential, so that steroids therapy can be started as soon as possible to prevent complications. Doppler ultrasonography of the temporal arteries provides rapid, non-invasive diagnostic support. However, the recommendations do not specify how soon temporal artery Doppler should be performed after steroids treatment, except that the halo sign would disappear after about 5 days on steroids. Sensitivity seems to be better when the examination is performed early, but the time taken for the halo sign to disappear is unknown. The investigator suggests that the disappearance of the temporal artery halo sign in GCA patients is observed earlier than D14 of steroids treatment usually reported in the literature. He speculates that the sensitivity of the temporal artery Doppler decreases as early as D3 of steroids treatment, and that beyond D7 it is not useful to perform this examination as its sensitivity becomes too low.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 and over
* Without legal protection.
* Meeting GCA classification criteria as defined by ACR 2022.
* Newly diagnosed with an indication for corticosteroid treatment.
* Have not yet received corticosteroid treatment for GCA.
* No contraindication to corticosteroid treatment.
* Person affiliated with or benefiting from a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination necessary for the research).

Exclusion Criteria:

* Patients with a relapse of Giant Cell Arteritis (GCA).
* Patients who have previously undergone a temporal artery biopsy (TAB), including for other reasons.
* Patients who have received oral corticosteroid treatment in the past month or are currently on corticosteroid therapy (excluding hydrocortisone or local corticosteroids).
* Patients with other types of vasculitis that may constitute a differential diagnosis: presence of antibodies against the cytoplasm of neutrophils (ANCA), positive syphilis serology, positivity of an IGRA test (Interferon Gamma Release Assay).
* Patients having received immunosuppressive treatment or biotherapy in the month prior to inclusion. If the patient's condition warrants the use of biotherapy or immunosuppressive treatment, its initiation will be delayed until after Day 7 to avoid interfering with the Doppler procedure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with GCA AND temporal artery Doppler WITH a halo sign on Day 0 of corticosteroid therapy and disappearing on Day 3. | From Day 0 to Day 3 of corticosteroid therapy

SECONDARY OUTCOMES:
Assessment of vasculitis via Doppler on Day 3, Day 7, and Day 15 | On Day 3, Day 7 and Day 15 of corticosteroid therapy
  With Doppler ultrasound, the following signs of vasculitis will be assessed : Difficulty compressing the temporal artery, Temporal artery occlusion, Temporal artery stenosis, Bilateral or unilateral halo sign and Presence of halo sign on vascular axes other than temporal arteries. The absence or presence of these signs will be reported and used to evaluate the disappearance of the halo sign over time during corticosteroid therapy.
Assessment of other vascular axes on Day 3 | On Day 3 of corticosteroid therapy
  Number of patients with positive echo-Doppler signs of vasculitis in subclavian, axillary, common/external/internal carotid and vertebral arteries.
Assessment of the number of patients with disappearance of the halo sign on Day 7 | On Day 7 of corticosteroid therapy
Assessment of the number of patients with disappearance of the halo sign on Day 15 | On Day 15 of corticosteroid therapy
Correlation between histological arteritis and echo-doppler halo sign | On Day 0 of corticosteroid therapy
  Number of patients with positive histology on temporal artery biopsy (to be performed at investigator's discretion)
Correlation between C-reactive protein (CRP) kinetics and disappearance of the halo sign | On Day 3 and Day 7 of corticosteroid therapy
  Number of patients with positive C-reactive protein (CRP) on Day 3 and Day 7
Correlation between corticosteroid dose and disappearance of halo sign | From Day 0 to Day 15
  * Number of patients receiving methylprednisolone bolus
  * Number of patients receiving prednisone equivalent greater than or equal to 60mg per day
Number of patients on Tocilizumab with disappearance of Halo sign on Day 15 | On Day 15 of corticosteroid therapy

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre Hospitalier du Mans, Le Mans, Sarthe
  - CHU d'Angers, Angers
  - CHU Caen Normandie, Caen
  - CHU Dijon - Hôpital François Mitterrand, Dijon
  - Groupe hospitalier La Rochelle-Ré-Aunis, La Rochelle
  - CHU Nantes, Nantes